CLINICAL TRIAL: NCT05683860
Title: A Multicenter, Open-label Extension (OLE) Study to Evaluate the Safety, Pharmacodynamics, and Clinical Effects of WVE-004 in Patients With C9orf72-associated Amyotrophic Lateral Sclerosis (ALS) and/or Frontotemporal Dementia (FTD)
Brief Title: Open-label Extension (OLE) Study of WVE-004 in Patients With C9orf72-associated Amyotrophic Lateral Sclerosis (ALS) and/or Frontotemporal Dementia (FTD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Despite robust, sustained reductions in poly(GP), no clinical benefit was seen at 24 weeks, and reductions in poly(GP) were not associated with stabilization in functional outcomes. Based on these data, Wave decided to stop development of WVE-004.
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVE-004-002
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-01

CONDITIONS: ALS; FTD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: WVE-004 (Dose A) (Experimental)
  Interventions: Drug: WVE-004

INTERVENTIONS:
Drug: WVE-004 — WVE-004 is a stereopure antisense oligonucleotide. It is administered via intrathecal injection

SUMMARY:
This is an OLE study conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and clinical effects of WVE-004 in adult patients with ALS, FTD, or mixed ALS/FTD phenotype with a documented mutation in the C9orf72 gene. To participate in the study, patients must have successfully completed Phase 1b/2a WVE-004-001 study.

ELIGIBILITY:
Inclusion Criteria:

* Patient successfully completed the Phase 1b/2a study with WVE-004, WVE-004-001.

Exclusion Criteria:

* Patient has a clinically significant medical finding on the physical examination other than C9orf72-associated ALS or FTD that, in the judgment of the Investigator or Sponsor, will make the patient unsuitable for participation in and/or completion of the trial procedures.
* Patient received any other investigational drug, biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Patient received an investigational oligonucleotide within the past 6 months or 5 half-lives of the drug, whichever is longer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety: Number of patients with adverse events (AEs) | Day 1 to Week 120 (end of study)
Safety: Number of patients with a severe AE | Day 1 to Week 120 (end of study)
Safety: Number of patients with serious AEs (SAEs) | Day 1 to Week 120 (end of study)
Safety: Number of patients who withdraw due to AEs | Day 1 to Week 120 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (3):
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- University of Oxford - Nuffield Department of Clinical Neurosciences, Oxford, United Kingdom